CLINICAL TRIAL: NCT02346253
Title: A Phase I/II Study of High-Dose-Rate Brachytherapy as Monotherapy for Prostate Cancer
Brief Title: High-Dose Brachytherapy in Treating Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-32058; NCI-2015-00089 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0065 (Other: OnCore)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; bicalutamide; Leuprolide; Goserelin; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (HDR brachytherapy, ADT and LHRH agonist therapy) (Experimental): Patients undergo high-dose-rate brachytherapy over 2 fractions. Patients also receive ADT comprising bicalutamide PO QD. Patients may also receive LHRH agonist therapy comprising leuprolide acetate IM or SC, goserelin acetate SC, triptorelin pamoate IM, or degarelix SC for 4-6 months (intermediate-risk patients receiving ADT) or 6-36 months (high-risk patients) at the discretion of the treating physician.
  Interventions: Radiation: Internal Radiation Therapy; Drug: Bicalutamide; Drug: Leuprolide Acetate; Drug: Goserelin Acetate; Drug: Triptorelin Pamoate; Drug: Degarelix; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Internal Radiation Therapy — Undergo high-dose-rate brachytherapy
  Other Names: Brachytherapy; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Drug: Bicalutamide — Given PO
  Other Names: CDX
Drug: Leuprolide Acetate — Given IM or SC
  Other Names: A-43818
Drug: Goserelin Acetate — Given SC
  Other Names: ICI-118630; ZDX; Zoladex
Drug: Triptorelin Pamoate — Given IM
  Other Names: Pamorelin; Trelstar
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies the side effects and how well high-dose brachytherapy works in treating patients with prostate cancer that has not spread to other parts of the body. Brachytherapy is a type of radiation therapy in which radioactive material sealed in needles, seeds, wires, or catheters is placed directly into or near a tumor and may be a better treatment in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To estimate the rate of acute (within 6 months of high-dose rate [HDR] completion) grade ≥ 2 genitourinary (GU) toxicity following high-dose-rate (HDR) brachytherapy (BT) as monotherapy for newly-diagnosed prostate cancer using the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 3 (CTCAE v3.0).

SECONDARY OBJECTIVES:

* Estimate the proportion of men with a prostate-specific antigen (PSA) nadir by one year (nPSA12) of < 2 ng/mL.
* Estimate the rate of freedom from biochemical failure at 5 years (FFBF).
* Evaluate patient-reported quality of life via the 32-item Expanded Prostate Cancer Index Composite (EPIC).
* Assess the cost-effectiveness of HDR BT as monotherapy for prostate cancer using the 6-item European Quality of Life 5-Dimensions (EQ-5D).
* Explore pre-treatment clinical risk factors to optimize patient selection for HDR BT as monotherapy for prostate cancer.
* Compare acute and late (> 6 months after HDR completion) GU and gastrointestinal (GI) grade ≥ 2 toxicity using CTCAE v3.0 and v4.0.
* Explore dosimetric predictors of toxicity.

Patients undergo high-dose-rate brachytherapy over 2 fractions. Patients may receive androgen deprivation therapy (ADT) comprising bicalutamide orally (PO) once daily (QD). Patients may also receive luteinizing hormone-releasing hormone (LHRH) agonist therapy comprising leuprolide acetate intramuscularly (IM) or subcutaneously (SC), goserelin acetate SC, triptorelin pamoate IM, or degarelix SC for 4 to 6 months (intermediate-risk patients receiving ADT) or 6 to 36 months (high-risk patients) at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months, and then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented pathologic confirmation of prostate adenocarcinoma
* Clinical T-classification T1-3
* PSA < 150 ng/mL
* Gleason score 6-10
* Clinically negative lymph nodes as established by abdomino-pelvic CT. CT only for clinical classification of T3 (with contrast if renal function is acceptable; a non-contrast CT is permitted if the patient is not a candidate for contrast), magnetic resonance imaging (MRI), nodal sampling, or dissection. Patients with lymph nodes equivocal or questionable by imaging are eligible if those nodes are <1 cm in short axis diameter. [56]
* No evidence of bone metastases (M0) on bone scan, only for PSA >20 ng/mLor Gleason ≥8, (NaF PET/CT is an acceptable substitute). Equivocal bone scan findings are allowed if plain films and/or MRI are negative for definite metastases.
* American Urological Association Symptom Index (AUA SI) =< 20

Exclusion Criteria:

* Clinical T4 disease
* PSA >= 150 ng/mL
* AUA SI > 20
* History of radical prostatectomy, external beam radiotherapy (EBRT), or BT for prostate cancer
* Previous chemotherapy for any malignancy, if given within three years of registration
* History of rectal surgery
* History of rectal fistula
* History of inflammatory bowel disease
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last six months
  * Transmural myocardial infarction within the last six months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with acute grade 2 or greater acute GU toxicity, scored according to CTCAE v3.0 | Within 6 months of HDR completion
  Will be calculated with a 90% confidence interval. Treatment plans will be reviewed, and doses to normal structures will be calculated and tabulated to determine possible relationships with toxicity outcomes.

SECONDARY OUTCOMES:
Proportion of men with a nPSA12 of < 2 ng/mL | Up to 1 year after completion of HDR
  nPSA12 is defined as the lowest PSA level achieved during the first year after completing HDR.
FFBF (Biochemical failure define according to PSA nadir+2ng/mL and 3 consecutive rises definition according to American Society of Radiation Oncology | From the completion of all treatment to the time of BF, assessed at 5 years
  Biochemical failure (BF) will be defined according the PSA nadir + 2 ng/mL and three consecutive rises definition according to the American Society of Radiation Oncology consensus recommendation. Time to first BF will be analyzed with competing risk models with death as a competing risk.
Change in quality of life as measured by EPIC scores | Baseline to up to 5 years
Cost-effectiveness of HDR BT as monotherapy for prostate cancer using as measured by EQ-5D scores | Up to 5 years
  Measured utility values for each patient on this study will be combined with overall survival to calculate the "QALY" quality-adjusted life years.
Pre-treatment clinical risk factors to optimize patient selection for HDR BT as monotherapy for prostate cancer (association between each risk factor and the risk of having a first BF) | Baseline
  Clinical risk factors will be tested in competing risk models to evaluate the association between each risk factor and the risk of having a first BF.
Proportion of patients with acute grade 2 or greater acute GU toxicity, scored according to CTCAE v4.0 | Within 6 months of HDR completion
  Will be calculated with a 90% confidence interval. Treatment plans will be reviewed, and doses to normal structures will be calculated and tabulated to determine possible relationships with toxicity outcomes.
Late GU toxicity, scored according to CTCAE v3.0 and v4.0 | Up to 5 years
  Will be calculated with a 90% confidence interval. Treatment plans will be reviewed, and doses to normal structures will be calculated and tabulated to determine possible relationships with toxicity outcomes.
Acute GI toxicity scored according to CTCAE v3.0 and CTCAE v4.0 | Up to 6 months after completing HDR BT
  Will be calculated with a 90% confidence interval. Treatment plans will be reviewed, and doses to normal structures will be calculated and tabulated to determine possible relationships with toxicity outcomes.
Late GI toxicity, scored according to CTCAE v3.0 and CTCAE v4.0 | Up to 5 years
  Will be calculated with a 90% confidence interval. Treatment plans will be reviewed, and doses to normal structures will be calculated and tabulated to determine possible relationships with toxicity outcomes.
Dosimetric predictors of toxicity (Doses to pelvic structures will be calculated and reviewed to determine possible correlations with toxicity outcomes) | Up to 5 years
  Doses to pelvic structures will be calculated and reviewed to determine possible correlations with toxicity outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Buyyounouski, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States